CLINICAL TRIAL: NCT01077037
Title: Impact of a Decision Aid on Patient Participation in Decision Making and Resource Use in Low Risk Chest Pain Patients: A Randomized Trial
Brief Title: Impact of a Decision Aid on Patient Decision Making in Emergency Department Chest Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erik P. Hess, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-006263
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Experimental): Receives Decision Aid
  Interventions: Other: Decision Aid
- Control (No Intervention): Patient receives usual care.

INTERVENTIONS:
Other: Decision Aid — Chest pain choice decision aid
  Arms: Decision Aid

SUMMARY:
We are doing a study to assess the impact of including patients in making decision regarding their own medical care in the emergency department. We will randomly assign them to either receive a decision aid or usual care. In doing this, we aim to increase patient satisfaction and safely decrease medical cost.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a primary complaint of chest pain.
* Treating clinician's next consideration is observation unit admission for cardiac stress testing.

Exclusion Criteria:

* Initial cardiac troponin T value >99th percentile (>0.01ng/mL)
* History of coronary artery disease
* coronary revascularization procedure within the previous 30 days
* cocaine use within 72 hours by the clinician's initial history
* pregnancy
* patient cannot read English or have, in their clinician's judgment, major learning barriers, such as visual or hearing impairment or dementia that would compromise their ability to give written informed consent (or use the decision aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Patient knowledge | Immediately after patient visit
  Patient knowledge regarding their short-term risk for an ACS and the risks of radiation exposure.

SECONDARY OUTCOMES:
Quality of decision making process | Immediately after patient visit
  Quality of the decision making process for the patient and clinician
Satisfaction with decision aid | Immediately after patient visit
  Patient and clinician acceptability and satisfaction with the decision aid
Proportion of patients who decided to undergo observation unit admission and urgent cardiac stress testing | During the initial ED visit
  Proportion of patients who decided to undergo observation unit admission and urgent cardiac stress testing
Delayed or missed ACS | 30 days
  Rate of delayed or missed ACS
Economic costs and healthcare utilization | 30 days
  Economic costs and healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Erik P Hess, MD, MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289
- [Derived] Izzo R, de Simone G, Trimarco V, Giudice R, De Marco M, Di Renzo G, De Luca N, Trimarco B. Primary prevention with statins and incident diabetes in hypertensive patients at high cardiovascular risk. Nutr Metab Cardiovasc Dis. 2013 Nov;23(11):1101-6. doi: 10.1016/j.numecd.2012.11.002. Epub 2013 Feb 15. PMID 23419735
- [Derived] Hess EP, Knoedler MA, Shah ND, Kline JA, Breslin M, Branda ME, Pencille LJ, Asplin BR, Nestler DM, Sadosty AT, Stiell IG, Ting HH, Montori VM. The chest pain choice decision aid: a randomized trial. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):251-9. doi: 10.1161/CIRCOUTCOMES.111.964791. Epub 2012 Apr 10. PMID 22496116
- [Derived] Pierce MA, Hess EP, Kline JA, Shah ND, Breslin M, Branda ME, Pencille LJ, Asplin BR, Nestler DM, Sadosty AT, Stiell IG, Ting HH, Montori VM. The Chest Pain Choice trial: a pilot randomized trial of a decision aid for patients with chest pain in the emergency department. Trials. 2010 May 17;11:57. doi: 10.1186/1745-6215-11-57. PMID 20478056